CLINICAL TRIAL: NCT07370831
Title: External Validation Study of a Laboratory-based Perioperative Prediction Model for Acute Kidney Injury After Cardiac Surgery.
Brief Title: Incidence and Prognostic of Cardiac Surgery-Associated Acute Kidney Injury: A Spanish Multicenter Study (SCARS-AKI)
Acronym: SCARS-AKI
Status: Completed | Type: Observational
Sponsor: Universidad de Oviedo (Other)
Responsible Party: Principal Investigator, Luis Baeza Álvarez, Principal Investigator, Universidad de Oviedo
Other Study IDs: CEImPA 2023.111
Record Dates: First submitted 2026-01-12; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Surgery Associated - Acute Kidney Injury; CKD (Chronic Kidney Disease) Stage 5D; Acute Kidney Injury; Acute Kidney Disease
Keywords: CSA AKI; AKI
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: CARDIAC SURGERY — PATIENTS UNDERGOING CARDIAC SURGERY

SUMMARY:
To predict the renal damage caused by cardiac surgery in patients to try to mitigate it as soon as possible

DETAILED DESCRIPTION:
Acute Kidney Injury (AKI) is a major complication of cardiac surgery and its most severe forms are associated with significant morbidity and mortality .

Identification of patients at risk may facilitate early use of management protocoolos recommended by KDIGO (Kidney Disease: Improving Global Outcomes), such as haemodynamic and volume optimisation, monitoring of renal function and discontinuation or reduction of nephrotoxic drugs . The rate associated with cardiac surgery varies according to its different historical definitions, from 0.3% to 29.7% . Cases requiring renal replacement therapy (RRT) occur between 1 .2%-3.0% in the studied cardiac surgery cohorts and their presence is a n independent predictor of mortality.

Because AKI still lacks effective treatments in addition to support and elimination of the cause, early and specific diagnosis is an unmet but critical need f o r successful and personalised patient management.

Creatinine, urea and urine output have been and are the main ways to diagnose and treat renal failure. Other types of biomarkers that seem to be related to risk of postoperative AKI are currently under study. Although more research is needed, they may eventually become predictive diagnostic tools. Several studies have indicated that the urinary level of NGAL excreted intraoperatively and after surgery is effective in predicting AKI in both adult and paediatric populations. Similar results have been obtained with other urinary biomarkers, such as the cell cycle arrest biomarkers TIMP-2 and IGFBP7) KIM-1, NAG, IL-18 and L-FAP . The major limitation of these biomarkers is that they are not easily accessible in all hospitals and clinical settings. Recently Demirjian developed a predictive model in which they observed that perioperative change in serum creatinine and postoperative blood urea nitrogen, serum sodium, potassium, bicarbonate and albumin from the first metabolic panel after cardiac surgery show good predictive value for moderate to severe AKI within 72 hours and 14 days after the surgical procedure.

3. Hypothesis

The score developed by Demirjian et al has a good predictive ability for moderate to severe AKI after cardiac surgery in the European population.

4. Objectives

4.1 Main

* Confirm the usefulness and externally validate the scale.
* Compare this scale with other models of AKI prediction after cardiac surgery: Thakar, Mehta, ISR, Callejas, Leicester, CRATE.

4.2 Secondary

* Identify new risk factors for Acute Kidney Injury (AKI)
* Understanding the incidence of AKI after cardiac surgery in Europe
* Validating a model for predicting discharge dialysis after cardiac surgery
* Investigate the performance of these models in specific surgeries: coronary surgery without cardiopulmonary bypass and heart transplantation.
* Assess the performance of other scales and compare them.
* Determine the prevalence and risk factors for Acute Kidney Disease (AKD) (renal injury beyond 7 days, up to 90 days).
* Determine the prevalence and risk factors for new Chronic Kidney Disease (CKD) (follow-up for 120 days or 4 months).
* Determine the prevalence and risk factors for CKD progression, defined by a one-stage progression in patients with pre-existing CKD. Follow-up for 120 days (4 months).

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age undergoing cardiac surgery.

Exclusion Criteria:

* Exitus in the first 48h postoperative period
* Patient undergoing renal replacement therapy or preoperative dialysis
* Minor" cardiac surgery ( sternal dehiscence, MCP removal or implantation, pericardial window)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years old undergoing all types of major cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
- Confirm the usefulness and externally validate the Demijirian scale. | up to 14th postoperative day
  Validate scale
- Compare this scale with other models of AKI prediction after cardiac surgery: Thakar, Mehta, ISR, Callejas, Leicester, CRATE. | up to 14th postoperative day
  Score validation

SECONDARY OUTCOMES:
- Identify new risk factors for Acute Kidney Injury (AKI) | from surgery to 4months postoperative
  AKI risk factor
- Validating a model for predicting discharge dialysis after cardiac surgery | from surgery to 4monts postoperative
  Develope a dialysis after cardiac surgery score
risk factors for new Chronic Kidney Disease (CKD) | from surgery to 4months postoperative
  Determine the prevalence and risk factors for new Chronic Kidney Disease (CKD) (follow-up for 120 days or 4 months).
Drugs related with CSA AKI | from surgery to 4months postoperative
  Study relation of : ISGLP2, GLP2, IDPP4, Sacubitril/valsartan with CS AKI

CONTACTS AND LOCATIONS:
Overall Officials: Luis Baeza Alvarez, MD, Principal Investigator — Universidad de Oviedo; Marc Vives Santacana, PhD, Study Director — Clinica Universidad de Navarra; Pablo Avanzas Fernández, PhD, Study Director — Universidad de Oviedo
Locations (1):
- HUCA, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No
Not necessary

REFERENCES:
- [Result] Demirjian S, Bashour CA, Shaw A, Schold JD, Simon J, Anthony D, Soltesz E, Gadegbeku CA. Predictive Accuracy of a Perioperative Laboratory Test-Based Prediction Model for Moderate to Severe Acute Kidney Injury After Cardiac Surgery. JAMA. 2022 Mar 8;327(10):956-964. doi: 10.1001/jama.2022.1751. PMID 35258532
- [Result] Mehta RH, Grab JD, O'Brien SM, Bridges CR, Gammie JS, Haan CK, Ferguson TB, Peterson ED; Society of Thoracic Surgeons National Cardiac Surgery Database Investigators. Bedside tool for predicting the risk of postoperative dialysis in patients undergoing cardiac surgery. Circulation. 2006 Nov 21;114(21):2208-16; quiz 2208. doi: 10.1161/CIRCULATIONAHA.106.635573. Epub 2006 Nov 6. PMID 17088458
- [Result] Lange HW, Aeppli DM, Brown DC. Survival of patients with acute renal failure requiring dialysis after open heart surgery: early prognostic indicators. Am Heart J. 1987 May;113(5):1138-43. doi: 10.1016/0002-8703(87)90925-2. PMID 3578008

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT07370831/Prot_SAP_000.pdf